CLINICAL TRIAL: NCT03726736
Title: Anlotinib Combined With Docetaxel Versus Docetaxel for Platinum-based Therapy Treated Advanced NSCLC: a Multicentre, Randomised Explorative Trial
Brief Title: Anlotinib Combined With Docetaxel Versus Docetaxel for Previous Treated Advanced NSCLC
Acronym: ACWDVDFPTAN
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yong Fang (Other)
Collaborators: Zhejiang Provincial People's Hospital (Other); Zhejiang Cancer Hospital (Other); Ningbo No. 1 Hospital (Other); Ningbo No.2 Hospital (Other); Affiliated Hospital of Jiaxing University (Other); Huzhou Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Yong Fang, professor, Sir Run Run Shaw Hospital
Organization: Sir Run Run Shaw Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L016
Record Dates: First submitted 2018-10-23; First posted 2018-10-31 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2018-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib combined Docetaxel (Experimental): patients treated with anlotinib and Docetaxel (21 days for 1 cycle) until PD (progressive disease)
  Interventions: Drug: Anlotinib combined Docetaxel
- Docetaxel (Active Comparator): patients treated with Docetaxel (21 days for 1 cycle) until PD (progressive disease)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Anlotinib combined Docetaxel — Anlotinib ( dose base on phase I study, QD PO d1-14, 21 days per cycle) and Docetaxel (60mg/m2 IV, d1, 21 days per cycle)
  Arms: Anlotinib combined Docetaxel
Drug: Docetaxel — Docetaxel (60mg/m2 IV, d1, 21 days per cycle)
  Arms: Docetaxel

SUMMARY:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor in domestic research and development. It can inhibit the angiogenesis related kinase, such as VEGFR, FGFR, PDGFR, and tumor cell proliferation related kinase -c-Kit kinase. In the phase Ⅲ study, patients who failed at least two kinds of systemic chemotherapy (third line or beyond) or drug intolerance were treated with anlotinib（12mg，po. qd. on day 1to14 of a 21-day cycle） or placebo, the anlotinib group PFS and OS were 5.37 months and 9.63 months, the placebo group PFS and OS were 1.4 months and 6.3 months. Therefore,we envisage using anlotinib plus docetaxel treat the EGFR wild-type advanced Non-small cell lung cancer patients who were failure in the treatment of chemotherapy with platinum containing drugs, to further improve the patient's PFS or OS.

DETAILED DESCRIPTION:
This multicentre randomised controlled clinical trial conducted in China include phase I study and phase II study.

Phase I study: to get the maximum tolerated dose of anlotinib when combined with Docetaxel.

Phase II study: to compare the effectiveness and safety of Anlotinib Plus Docetaxel in patients of EGFR wild-type Advanced Non-squamous Non-small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects voluntarily joined the study and signed informed consent, with good compliance and follow-up;
* 2. Diagnosed as locally advanced and / or metastatic non-small cell lung adenocarcinoma (NSCLC) by cytology or histology; diagnosed as stage IIIB, IIIC or IV according to the 2017 new version of the UICC lung cancer staging criteria (8th edition);
* 3. At least one target lesion that has not received local treatment in the past 3 months, and accurate measurement by magnetic resonance imaging (MRI) or computed tomography (CT) in at least 1 direction
* 4. first line chemotherapy used platinum-based doublet chemotherapy and failed.
* 5. Provide detectable specimens (tissue or cancerous pleural effusion) for genotyping before enrollment, and the patients should be with negative EGFR, ALK, and ROS1 gene test results;
* 6. 18~75 years old, ECOG PS 0-1 points. Life expectancy is at least 3 months.
* 7. The damage subjects received from other treatments has recovered(NCI-CTCAE version 4.0 grade ≤ 1), the interval of subjects receiving nitrosourea or mitomycin should be at least 6 weeks; the interval subjects receiving other cytotoxic drugs, bevacate Avastin (Avastin), surgery should be at least 4 weeks; the interval subjects receiving radiotherapy (except for local palliative radiotherapy) should be at least 2 weeks;
* 8. The main organs function are normally, the following criteria are met:

  1. Blood routine examination criteria should be met (no blood transfusion and blood products within 14 days, no correction by G-CSF and other hematopoietic stimuli): HB≥90 g/L; ANC ≥ 1.5×10^9/L; PLT ≥80×10^9/L;
  2. Biochemical examinations must meet the following criteria: TBIL<1.5×ULN; ALT and AST < 2.5×ULN, and for patients with liver metastases < 5×ULN; Serum Cr ≤ 1.25×ULN or endogenous creatinine clearance > 60 ml/min (Cockcroft-Gault formula).
* 9. Avoid pregnancy during treatment and 6 month after treatment.

Exclusion Criteria:

* 1. Small cell lung cancer (including lung cancer mixed with small cell lung cancer and non-small cell lung cancer);
* 2. Have used anlotinib / docetaxel before, or have used other VEGFR-TKI drugs.
* 3. Imaging (CT or MRI) shows that the distance between tumor lesion and the large blood vessel is ≤ 5 mm, or there is a central tumor that invades the local large blood vessel; or there is a significant pulmonary cavity or necrotizing tumor;
* 4. History and comorbidities

  1. Active brain metastases, cancerous meningitis, spinal cord compression, or imaging CT or MRI screening for brain or pia mater disease (a patient with brain metastases who have completed treatment and stable symptoms in 28 days before enrollment may be enrolled, but should be confirmed by brain MRI, CT or venography evaluation as no cerebral hemorrhage symptoms);
  2. The patient is participating in other clinical studies or completing the previous clinical study in less than 4 weeks;
  3. Other active malignancies that require simultaneous treatment;
  4. Patients with a history of malignant tumors except for patients with cutaneous basal cell carcinoma, superficial bladder cancer, cutaneous squamous cell carcinoma or orthotopic cervical cancer who have undergone a curative treatment and have no disease recurrence within 5 years from the start of treatment
  5. Patients with previous anti-tumor treatment-related adverse reactions (excluding hair loss) who have not recovered to NCI-CTCAE ≤1;
  6. Abnormal blood coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy;
  7. Note: Under the premise of prothrombin time international normalized ratio (INR) ≤ 1.5, low-dose heparin (adult daily dose of 0.6 million to 12,000 U) or low-dose aspirin (daily dosage ≤ 100 mg) is allowed for preventive purposes;
  8. Renal insufficiency: urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0g;
  9. Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite optimal medical treatment);
  10. The effects of surgery or trauma have been eliminated for less than 14 days before enrollment in subjects who have undergone major surgery or have severe trauma;
  11. Severe acute or chronic infections requiring systemic treatment;
  12. Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including men with QTc interval ≥ 450 ms, women ≥ 470 ms); according to NYHA criteria, grades III to IV Insufficient function, or cardiac color Doppler ultrasound examination indicates left ventricular ejection fraction (LVEF) <50%;
  13. There is currently a peripheral neuropathy of ≥CTCAE 2 degrees, except for trauma;
  14. Respiratory syndrome (≥CTC AE grade 2 dyspnea), serous effusion (including pleural effusion, ascites, pericardial effusion) requiring surgical treatment;
  15. Long-term unhealed wounds or fractures;
  16. Severe weight loss (greater than 10%) within 6 weeks prior to randomization;
  17. Decompensated diabetes or other ailments treated with high doses of glucocorticoids;
  18. Factors that have a significant impact on oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
  19. Clinically significant hemoptysis (daily hemoptysis greater than 50ml) within 3 months prior to enrollment; or significant clinically significant bleeding symptoms or defined bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ and above, or suffering from vasculitis;
  20. Events of venous/venous thrombosis occurring within the first 12 months prior to enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
  21. Planned for systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (4 weeks prior to enrollment in other anti-cancer drug clinical trials or within 4 weeks prior to grouping or during the study period Or use mitomycin C) within 6 weeks prior to receiving the test drug. Radiation-rehabilitation radiotherapy (EF-RT) was performed within 4 weeks before grouping or limited-field radiotherapy to be evaluated for tumor lesions within 2 weeks before grouping.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
PFS | each 42 days up to PD or death(up to 24 months)
  Progress free survival

SECONDARY OUTCOMES:
OS | From randomization until death (up to 24 months)
  Overall Survival
quality of life | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  use EORTC QLQ-C30(version 3) questionnaire to evaluate the quality of life
ORR | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Objective Response Rate
DCR | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Disease Control Rate
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Until 21 day safety follow-up visit
  Record Adverse Events (AEs) according to CTCAE (V4.03). To find Potential adverse reaction, measure blood pressure at least 2 times a week and test blood routine, Blood biochemical, Urine routine, stool routine, coagulation function, electrocardiogram for each follow-up, record and analyze the number of abnormal data.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shou J, Chen J, Guo Q, Hong W, Wang Y, Rao C, Lu L, Yang X, Zhu D, Lan F, Fang Y, Pan H. Anlotinib in combination with docetaxel for advanced nonsmall cell lung cancer after failure of platinum-based treatment: A phase 1/2 trial. Cancer. 2025 May 15;131(10):e35822. doi: 10.1002/cncr.35822. PMID 40366884
- [Derived] Pu X, Shou J, Xiao Z, Chen J, Xiao M, Guo Q, Ma Z, Hong W, Wang Q, Wang Y, Li J, Rao C, Weng J, Lu L, Wu L, Fang Y. Anlotinib Plus Docetaxel is Promising in Advanced NSCLC Progressing on First-Line Immunotherapy: A Pooled Analysis of Two Randomized Trials. Adv Ther. 2025 Jul;42(7):3249-3264. doi: 10.1007/s12325-025-03170-2. Epub 2025 May 12. PMID 40354010